CLINICAL TRIAL: NCT05750030
Title: Fecal Microbiota Transplant (FMT) Combined With Atezolizumab Plus Bevacizumab in Patients With HepatoCellular Carcinoma Who Failed to Respond to Prior Immunotherapy - the FAB-HCC Pilot Study
Brief Title: FMT in IT-refractory HCC - FAB-HCC Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Matthias Pinter, Clinical professor and principal investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAB0001; 2022-000234-42 (EudraCT Number)
Record Dates: First submitted 2023-01-16; First posted 2023-03-01 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Fecal Microbiota Transplant; Hepatocellular Carcinoma; FMT; HCC; Immunotherapy; Atezolizumab; Bevacizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: 12 Patients with HCC who failed to achieve or maintain a complete or partial response (according to mRECIST) to atezolizumab plus bevacizumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FMT combined with Atezolizumab plus Bevacizumab (Experimental)
  Interventions: Combination Product: FMT combined with Atezolizumab plus Bevacizumab

INTERVENTIONS:
Combination Product: FMT combined with Atezolizumab plus Bevacizumab — Single FMT from patients with HCC who responded to PD-(L)1-based immunotherapy to patients with HCC who failed to achieve complete or partial response (according to mRECIST) to atezolizumab/bevacizumab. After single FMT, patients will continue to receive atezolizumab/bevacizumab every 21-days according to protocol.

SUMMARY:
This single-center, pilot study (phase IIa) will evaluate the safety, feasibility, and efficacy of FMT from patients with HCC who responded to PD-(L)1-based immunotherapy to patients with HCC who failed to respond to atezolizumab/bevacizumab.

DETAILED DESCRIPTION:
The main purpose of this phase IIa pilot study is to test the safety and efficacy of fecal microbiota transplant (FMT) combined with atezolizumab plus bevacizumab in patients who failed to achieve or maintain a complete or partial radiological response (according to mRECIST) to prior immunotherapy for advanced hepatocellular carcinoma (aHCC).

The primary objective is to assess the safety of FMT combined with atezolizumab plus bevacizumab, as measured by incidence and severity of treatment-related adverse events.

The secondary objectives are to assess the efficacy of FMT in combination with atezolizumab plus bevacizumab as measured by best radiological response, objective response rate (ORR), disease control rate (DCR), progression-free survival (PFS), and overall survival (OS). Furthermore, the objective is to evaluate the impact of FMT with atezolizumab plus bevacizumab on the quality of life, as assessed by EQ-5D-5L questionnaires.

Finally, this study also aims to assess the following exploratory endpoints:

* the effect of FMT on recipient gut microbiota composition, diversity, rate of change from baseline, and similarity to donor stool composition over time (compared between responders and non-responders)
* the effect of FMT on immune activity in the gut
* metagenome assemblies and functional profiling before and after FMT
* single cell analyses of circulating immune cells before and after FMT
* serum and stool metabolomic and lipidomic signatures before and after FMT

This is a phase II, single-center, open-label pilot study. Twelve patients suffering from advanced-stage hepatocellular carcinoma will be enrolled in this trial. The planned duration for this study are 48 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Age ≥ 18 years
* Histologically or radiologically confirmed HCC
* Patients with progressive disease (according to mRECIST) during treatment with atezolizumab/bevacizumab (without or with prior complete or partial response as best radiological response according to mRECIST) OR patients with stable disease as best radiological response (according to mRECIST) after the first 12 months of atezolizumab/bevacizumab treatment
* Negative HIV test
* Patients with chronic hepatitis B must be under antiviral treatment and hepatitis B DNA must be < 500 IU/mL
* Variceal status must be known and if present, adequate medical or endoscopic treatment is required
* ECOG Performance Status 0-1
* Child-Pugh class A-B8
* Adequate hematological and end-organ function, defined as follows:
* AST and ALT < 10 x ULN
* Serum bilirubin < 3.5 mg/dL
* Albumin ≥ 28 g/L
* Serum creatinine ≤ 1.5 mg/dL
* Hemoglobin ≥ 8 mg/dL
* Platelet count ≥ 50 G/L
* Leukocytes ≥ 2.5 G/L
* Patients not receiving therapeutic anticoagulation: INR ≤ 2.3 or thromboplastin time ≥ 40%
* Women of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods
* Men must agree to remain abstinent (refrain from heterosexual intercourse) or use a condom

Exclusion Criteria:

* Known fibrolamellar carcinoma or mixed cholangiocellular carcinoma
* Massive tumor progression (> 100% increase in target lesions or progression associated with significant clinical deterioration)
* Uncontrolled ascites
* Overt hepatic encephalopathy or concomitant treatment with rifaximin
* Prior allogeneic stem cell or solid organ transplantation
* Active or history of severe autoimmune disease
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to study inclusion or unstable angina
* Severe infection within 4 weeks prior to study inclusion
* Pregnant or breastfeeding women
* Treatment with systemic immunosuppressive medication with the following exceptions:
* Acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for contrast allergy)
* Mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease or asthma, or low-dose corticosteroids for adrenal insufficiency
* Significant vascular disease (e.g., peripheral arterial thrombosis) within 6 months prior to study inclusion
* Major surgery within 4 weeks prior to study inclusion or minor surgery (excluding placement of a vascular access device) within 3 days prior to study inclusion
* History of gastrointestinal fistula or perforation, or intraabdominal abscess within 6 months prior to study inclusion
* Serious, non-healing wound or active ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Safety of atezolizumab/bevacizumab in combination with FMT, measured by incidence and severity of treatment-related adverse events, determined according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v.5.0. | 24 months

SECONDARY OUTCOMES:
Efficacy assessed by the number of study participants achieving complete response (CR), partial response (PR), stable disease (SD) or progressive disease (PD) as best radiological response evaluated according to mRECIST/ RECIST v1.1 criteria. | 24 months
Efficacy as assessed by objective response rate (ORR) and disease control rate (DCR). Objective response is defined as either complete or partial response, while disease control rate comprises complete/partial response as well as stable disease. | 24 months
Efficacy as assessed by progression-free survival (PFS) and overall survival (OS). | 24 months
Quality of life (QoL) as assessed by the patient-reported outcome EQ-5D-5L (European Quality of Life 5 Dimensions 3 Level Version) questionnaire. | 24 months

OTHER OUTCOMES:
Effect of FMT on recipient gut microbiota composition, diversity (alpha and beta), rate of change from baseline and similarity to donor stool composition over time as well as comparison of responders and non-responders. | 24 months
Effect of FMT on immune activity in the gut by analyzing gut tissue samples with immunohistochemistry staining of immune cells of patients receiving FMT. | 24 months
Differences in metagenome assemblies and functional profiling using shotgun metagenomic analysis of donor and recipient stool samples before and after FMT. | 24 months
Differences in single cell analyses of circulating immune cells in patients before and after FMT. | 24 months
Differences in serum and stool metabolomic and lipidomic signatures in patients before and after FMT. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Pinter, MD PhD, Principal Investigator — Medical University of Vienna, Internal Medicine III, Department of Gastroenterology and Hepatology
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Pomej K, Frick A, Scheiner B, Balcar L, Pajancic L, Klotz A, Kreuter A, Lampichler K, Regnat K, Zinober K, Trauner M, Tamandl D, Gasche C, Pinter M. Study protocol: Fecal Microbiota Transplant combined with Atezolizumab/Bevacizumab in Patients with Hepatocellular Carcinoma who failed to achieve or maintain objective response to Atezolizumab/Bevacizumab - the FAB-HCC pilot study. PLoS One. 2025 Apr 15;20(4):e0321189. doi: 10.1371/journal.pone.0321189. eCollection 2025. PMID 40233040